CLINICAL TRIAL: NCT02144727
Title: A Multicenter Randomized Clinical Trial of D1+ Versus D2 Distal Gastrectomy for Stage IB & II Advanced Gastric Cancer
Brief Title: A Clinical Trial of D1+ Versus D2 Distal Gastrectomy for Stage IB & II Advanced Gastric Cancer
Acronym: ADDICT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Young-Woo Kim, Head of Gastric Cancer Branch, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-13-712
Record Dates: First submitted 2014-03-04; First posted 2014-05-22 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D2 distal subtotal gastrectomy (Active Comparator): D2 distal subtotal gastrectomy D2 includes Nos.1.3,4sb,4d,5,6,7,8a,9,11p,and 12a nodes in Japanese classification. Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy
  Interventions: Procedure: D2 distal subtotal gastrectomy
- D1+ distal subtotal gastrectomy (Experimental): D1+ distal subtotal gastrectomy D1+ includes Nos.1,3,4sb,4d,5,6,7,8a,and 9 nodes in Japanese classification. Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy
  Interventions: Procedure: D1+ distal subtotal gastrectomy

INTERVENTIONS:
Procedure: D2 distal subtotal gastrectomy — D2 includes Nos.1.3,4sb,4d,5,6,7,8a,9,11p,and 12a nodes in Japanese classification. Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy.
  Arms: D2 distal subtotal gastrectomy
Procedure: D1+ distal subtotal gastrectomy — D1+ includes Nos.1,3,4sb,4d,5,6,7,8a,and 9 nodes in Japanese classification. Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy
  Arms: D1+ distal subtotal gastrectomy

SUMMARY:
In oncological aspect, D1+ lymph node dissection would be enough for early stage gastric cancer in advanced gastric cancer (stage IB/IIA/IIB ).

DETAILED DESCRIPTION:
■ Background of Hypothesis A. JCOG (Japanese Clinical Oncology Group) 9501 Study

: Addition of aorta lymph node dissection to D2 lymph node dissection does not increase survival rate.

Wide range of operation is not always the best treatment. If invasion rate can be kept as minimal as possible while maintaining survival rate, it can lead to more secure operation while also reducing the frequency of complication after the surgery. 20 It may be advantageous for patients in terms of operation time, cost, and quality of life.

B. COACT 1001 study A previous study which compared the feasibility of lymph node dissection in open surgery and lapraroscopic surgery for advanced gastric cancer.

11p, 12a lymph node (D2) resection rate: 79.2% and 88.8% respectively in all advance gastric cancer.

11p, 12a lymph node (D2) metastasis rate: 1.9% and 2.9% respectively. Subgroup analysis 11p, 12a lymph node resection in cStage IB/IIA: 74.5-80.0% and 86.7-96.1% respectively. : 0% metastasis rate for both.

lymph node dissection in cStage IIB/IIIA: 81.1-82.3% and 87.5-89.2% respectively.: metastasis rates are 2.1% and 2.4-12.1% respectively.

Application: 11p and 12a lymph nodes, which belong in D2 lymph nodes, need to be resected in advance gastric cancer in IIB stage or higher. However, in earlier stages of advance gastric cancer, the probability of metastasis is very low; therefore, resection of D1+ lymph nodes, excluding 11p and 12a, is enough.

ELIGIBILITY:
Inclusion Criteria :

* Histologically proven primary gastric adenocarcinoma
* T1N1, T2N0, T2N1, T3N0, T3N1 by CT scan (AJCC 7th classification) and intraoperative surgical staging prior to resectional procedure
* Location of primary tumor; antrum, or angle, lower body or mid body of the stomach
* No evidence of other distant metastasis
* Aged ≥ 20 year old
* Performance status (PS) of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale
* No prior treatment of chemotherapy or radiation therapy against any other malignancies, and no prior treatment for gastric cancer including endoscopic mucosal resection
* Adequate organ functions defined as indicated below:

  * WBC 3000/mm3 - 12,000/mm3
  * >serum Hemoglobin 8.0 g/dl
  * > serum Platelet 100 000/mm3
  * < serum AST 100 IU/l
  * <serum ALT 100 IU/l
  * < Total Bilirubin 2.0 mg/dl
* Written signed informed consent

Exclusion Criteria :

* Active double cancer (synchronous double cancer and metachronous double cancer within five disease-free years), excluding carcinoma in situ (lesions equal to intraepithelial or intramucosal cancer)
* Gastric remnant cancer
* ≥T4a in surgical staging before resection
* N2 or more (number of metastatic lymph nodes ≥3) in CT scan
* Histologically rare variants in WHO Classification such as Adenosquamous, Hepatoid, Squamous cell, Undifferentiated, , neuroendocrine carcinoma and others
* Pregnant or breast-feeding women
* Mental disorder(diagnosed with mental disorder on medical record)
* systemic administration of corticosteroids(include Herbal Medication)
* unstable angina or myocardial infarction within 6 months of the trial
* unstable hypertension
* severe respiratory disease requiring continuous oxygen therapy
* previous upper abdominal surgery except laparoscopic cholecystectomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1880 (Estimated)
Dates: Start 2014-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 year
  To test non-inferiority of survival of D1+ gastrectomy versus D2 gastrectomy for clinical stage I B & II advanced gastric cancer

SECONDARY OUTCOMES:
disease free survival | 3 year
  3 year disease free survival
Subgroup analysis of Laparoscopic surgery versus open surgery | 3 year , 5 year
  Subgroup analysis of Laparoscopic surgery versus open surgery in terms of 3 year relapse free survival and 5 year overall survival
Operating time | op day
  Operating time
Early postoperative complications | within 30 days
  Early postoperative complications
Long term postoperative complications | after 30 days
  Long term postoperative complications
Quality of life of the patients in terms of European quality of life questionnaire (EQ-5D) | baseline, 1 week, 1month, 6 month, 1 year, 3 year
  Quality of life of the patients in terms of European quality of life questionnaire (EQ-5D)
Overall cost for the treatment | operation day to discharge
  Overall cost for the treatment (from operative day to discharge day)
Finding biomarkers predicting lymph node metastasis and recurrence | 3 year
  Finding biomarkers predicting lymph node metastasis and recurrence for prediction of lymph node metastasis and recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Young Woo Kim, PhD, Principal Investigator — National Cancer Center, Korea
Locations (50):
- South Korea (50):
  - Kosin University Gospel Hospital, Busan, Busan
  - Pusan National University Hospital, Busan, Busan
  - Dong-A University Hospital, Busan, Busan
  - Dongnam Inst. Of Radiological & Medical Sciences, Busan, Busan
  - Inje University Haeundae Paik Hospital, Busan, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan, Chuncheongnam-Do
  - Keimyung University Dongsan Medical Center, Daegu, Daegu
  - Kyungpook National University Hospital, Daegu, Daegu
  - Kungpook National University Hospital, Daegu, Daegu
  - Daegu Veterans Hospital, Daegu, Daegu
  - Yeungnam University Medical Center, Daegu, Daegu
  - Daegu Catholic Univ. Medical Center, Daegu, Daegu
  - Chungnam National University Hospital, Daejeon, Daejeon
  - Konyang University Hospital, Metropolitan City Daejon, Daejon
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Dongguk University Medical Center, Goyang-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - The Catholic University of Korea St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Dongguk University Gyeongju Hospital, Gyeongju, Gyeongsangbuk-do
  - Gyengsang National University Hospital, Jinjoo, Gyeongsangnam-do
  - National Cancer Center, Goyang, Gyunggi-Do
  - Inha University Hospital, Incheon, Incheon
  - The Catholic University of Korea Incheon St. Mary's Hospital, Incheon, Incheon
  - Gachon University Gill Medical Center, Incheon, Incheon
  - Jeju National University Hospital, Jeju City, Jeju Special Self-Governing Province
  - Chonbuk National University Hospital, Jeonju, Jellabuk-Do
  - Chosun University Hospital, Gwangju, Jellanam-Do
  - Chonnam National University Hwasun Hospital, Hwasun-Gun, Jellanam-Do
  - Seoul National University Hospital, Seoul, Seoul
  - Seoul Red Cross Hospital, Seoul, Seoul
  - Severance Hospital, Seoul, Seoul
  - KyungHee University Medical Center, Seoul, Seoul
  - Hanyang University Medical Center, Seoul, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul, Seoul
  - VHS Medical Center, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Gangnam Severance Hospital, Seoul, Seoul
  - Korea University Anam Hospital, Seoul, Seoul
  - The Catholic University of Korea St. Mary's Hospital, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Korea Cancer Center Hospital, Seoul, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul, Seoul
  - Konkuk University Medical Center, Seoul, Seoul
  - Hallym University Sacred Heart Hospital, Seoul, Seoul
  - Korea University Guro Hospital, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul
  - Chung-Ang University Hospital, Seoul, Seoul
  - Ewha Womans University Medical Center, Seoul, Seoul